CLINICAL TRIAL: NCT01384279
Title: The Therapeutic Effects of Topiramate and Metformin on Second Generation Antipsychotics-induced Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beitou Armed Forces Hospital, Taipei, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuo-Tung Chiang, Beitou Armed Forces Hospital, Beitou Armed Forces Hospital, Taipei, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-099-03
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Obesity
Keywords: metformin; topiramate; obesity; metabolic syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Metformin; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- metformin, topiramate (Experimental)
  Interventions: Drug: metformin, topiramate

INTERVENTIONS:
Drug: metformin, topiramate — metformin 250 mg/d is gradually increased to 1000 mg/d over four weeks, and topiramate 50 mg/d is gradually increased to 200 mg/d over four weeks

SUMMARY:
The primary aim of the study is to investigate the efficacy of metformin and topiramate on second-generation antipsychotic-induced obesity. The secondary domain we look at is the adverse effects of both drugs. The investigators hypothesize that metformin and topiramate are effective in treating obesity induced by second-generation antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: schizophrenia or schizoaffective disorder
2. Age: 20 to 65
3. BMI>27
4. Receiving second-generation antipsychotics(Olanzapine, Clozapine, Quetiapine, Risperidone, Amisulpride, Zotepine)

Exclusion Criteria:

1. Allergy to metformin or topiramate
2. Currently taking metformin or topiramate
3. Currently taking drugs that may interact with topiramate, including carbamazepine, eslicarbazepine, oxcarbazepine, phenobarbital, phenytoin, primidone, amitriptyline, lithium, metformin, propranolol, and sumatriptan.
4. Being pregnant or planning to become pregnant during the study period,
5. History of hypertension, DM, liver or renal function impairment, cardiovascular disease, CVA, or neurological disorders
6. History of hypoglycemia
7. History of suicidal attempt
8. Current scale of Hamilton Depression Rating Scale>8

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The changes in metabolic panel as the primary outcome | up to six months
  Metabolic panel, which includes HDL-C, VLDL, LDL, cholesterol, triglycerides, insulin, leptin, BW, Glucose, blood pressure, and weight(with waist circumference and BMI) will be assessed every month

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (including psychiatric adverse events) as a Measure of Safety and Tolerability | up to six months
  We use Positive and Negative Syndrome Scale, the Hamilton Depression Rating Scale, clinical golbal impression-severity, and the Udvalg for Kliniske Undersøgelser Side Effect Rating Scale every month to investigate the participants' safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Chiang Kuo-Tung, M.D., Principal Investigator — Department of Psychiatry, Beitou Armed Forces Hospital, Taipei, Taiwan
Locations (1):
- Beitou Armed Forces Hospital, Taipei, Taiwan